CLINICAL TRIAL: NCT02607345
Title: 25gr. Glucomedics vs 25gr. Zusto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bart Keymeulen (Other)
Responsible Party: Sponsor-Investigator, Bart Keymeulen, MD PhD, AZ-VUB
Organization: AZ-VUB (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015/030
Record Dates: First submitted 2015-10-12; First posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucomedics® (Active Comparator): 25gr Glucomedics®
  Interventions: Dietary Supplement: Glucomedics®
- Zusto® (Experimental): 25gr Zusto®
  Interventions: Dietary Supplement: Zusto

INTERVENTIONS:
Dietary Supplement: Zusto — 25gr
  Arms: Zusto®
Dietary Supplement: Glucomedics® — 25gr
  Arms: Glucomedics®

SUMMARY:
Objective: to compare blood glucose and insulin responses after consumption of 100ml water, sweetened with 25gr Zusto® and 100ml water sweetened with 25gr Glucomedics® (standard drink)

DETAILED DESCRIPTION:
This is an experimental study enrolling 10 healthy female subjects. The study compares the blood glucose and insulin responses after consumption of 100ml water, sweetened with 25gr Zusto® and 100ml water sweetened with 25gr Glucomedics® (standard drink). Subjects need to be fasted for at least 8 hours before all visits. At visit 1, five women will consume the solution with 25gr Zusto®, the other five will have the solution with 25gr Glucomedics®. On visit 2, groups will be switched. Visit 1 and 2 will be performed within approximately one week interval.

Both drinks will be identical in amount of water and only be different by the use of 25gr Glucomedics® and 25gr Zusto®.

Before intake of the drink, vital signs, weight and bedside blood glucose and baseline blood samples - 15' and 0' for glucose, insulin and C-peptide will be taken at visit 1 and 2. Both drinks will be consumed within 5 minutes and time of start and end of intake of Zusto® / Glucomedics® will be documented.

Blood samples for glucose, insulin and C-peptide will be taken at 15', 30', 60', 90', 120' and 180' after start of intake 25gr Zusto® and 25gr Glucomedics®.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects
* Age between 30 and 50 years
* BMI between 20 and 30 kg/m²

Exclusion Criteria:

* No first degree relatives with mellitus type 1 or type 2
* No intake of medication with influence blood glucose levels
* Pregnant, breast feeding or planning to become pregnant during the study
* Employer of the investigator or study center with direct involvement in the proposed study or other studies under the direction of the investigator or study center

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
the difference in glycemic index between 25gr. Zusto® and 25gr. Glucomedics® | 1 month
  GI values will be calculated using the iAUC of Zusto® intake and Glucomedics® intake.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Keymeulen, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel

REFERENCES:
- [Derived] Pen JJ, Khorosheva G, Van de Velde U, Debroye C, Huyghebaert A, Rottiers R, Keymeulen B. Zusto: A new sweetening agent with low glycemic index. Clin Nutr ESPEN. 2018 Feb;23:103-106. doi: 10.1016/j.clnesp.2017.11.009. Epub 2017 Dec 7. PMID 29460783